CLINICAL TRIAL: NCT04132661
Title: A Phase IV, Crossover, Randomized, Double Blind and Placebo-controlled Clinical Trial to Evaluate the Mode of Action of a Single Dose of Bisacodyl in Subjects With Occasional Constipation
Brief Title: MRI Assessment of Mode of Action of Bisacodyl, Single Dose
Acronym: MODS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Robin Spiller, Professor of Gastroenterology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CHC-2019-12564
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Bisacodyl

STUDY DESIGN:
Intervention Model Description: Phase IV, single center, double blind, randomized (1:1 ratio), two arms (bisacodyl and placebo), single-dose, and crossover clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study is a double blind study with a randomization ratio 1:1. The subjects, the investigator and the Sanofi team will be blinded to the treatment sequences allocation until the database lock. The medicinal product and placebo are indistinguishable using exactly the same packing and form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bisacodyl (Experimental): 5 mg bisacodyl, one tablet once
  Interventions: Drug: Bisacodyl 5 milligram
- placebo (Placebo Comparator): placebo, one tablet once
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Bisacodyl 5 milligram — one single dose
  Other Names: dulcolax
  Arms: bisacodyl
Drug: Placebo oral tablet — one single dose
  Arms: placebo

SUMMARY:
Constipation remains an important unmet medical need. Patients are currently often dissatisfied with treatment, because of lack of predictability of the laxative, side effects (mainly abdominal pain) and perceived decrease of efficacy with time. A recent systematic review of a range of laxatives reported that bisacodyl increases the number of complete spontaneous bowel movements statistically significant compared to placebo. Recently non-invasive Magnetic Resonance Imaging (MRI) techniques have been developed to assess small intestinal fluid distribution, transit and motility as well as colonic fluid, volumes and motility in healthy volunteers and constipated subjects. Other laxatives such as movecol and ispaghula have been investigated using this methodology. This study will use these novel techniques to further characterize bisacodyl's mode of action.

This study is intended to assess the effect of a single-dose of bisacodyl on the gut motor function and its effect on water distribution within the small and large intestine in subjects with occasional constipation by MRI. It may allow better understanding of the relative importance of both the secretory and the prokinetic effect of bisacodyl.

Since bisacodyl is often used by self-medicating people with constipation it is proposed to study subjects suffering from occasional constipation. As such subjects often take the drug intermittently it would be of interest to study both the acute response after single dose and the response after several days of treatment to see if this alters the response.

The current study will be performed as a cross-over with 2-period and 2-treatment (bisacodyl/placebo), for assessing the effects over of a single-dose of 5mg bisacodyl.

Evaluations will be performed after one single dose of bisacodyl or placebo in two different time periods, separated by a 2 week washout period between end of period 1 and start of period 2.

The study will recruit individuals ≥18yrs from the general public who consider themselves as suffering from occasional constipation and who self-medicate with an occasional over-the counter (OTC) laxative, not more than once a week. Up to 18 adult healthy subjects will be recruited to ensure 10 evaluable subjects. An evaluable subject is defined as participant having the primary endpoint assessed (ascending colon T1 300, 375, and 450 minutes correctly evaluated) for the two periods of the crossover.

ELIGIBILITY:
Inclusion Criteria:

I 01. Adult subjects that self-medicate with occasional laxative no more than 4 times in the month before eligibility confirmation

I 02. Meet Rome IV criteria for Chronic Constipation.

I 03. ≥18 years of age inclusive, at the time of signing the informed consent.

I 04. Screening diary confirms they experience at least 2 days in the 7 day diary with either hard stools (Bristol Stool form Score 1 or 2) or no bowel movement

I 05. BMI under or equal to 35 kg/m2

I 06. Female subjects of child bearing potential must have a negative urine pregnancy test at screening. Subjects of child bearing potential or with partners of child bearing potential must agree to use methods of medically acceptable forms of contraception during the study and for 90 days after completion of study drug, (e.g. implants, injectable, combined oral contraceptives, barrier methods, true abstinence (when this is in line with the preferred and usual lifestyle of the patient) or vasectomised partners).

I 07. Capable of giving signed informed consent as described in Appendix 1 (Section 10.1) which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

E 01. Known hypersensitivity or other contraindications to bisacodyl use: such as ileus, intestinal obstruction, acute abdominal conditions including appendicitis, acute inflammatory bowel diseases, and severe abdominal pain associated with nausea and vomiting; and severe dehydration or rare hereditary conditions that may be incompatible with an excipient of the product (galactose intolerance, e.g. galactosaemia, fructose intolerance.

E 02. Pregnancy and/or breast breast-feeding or positive urine pregnancy test History of known gastrointestinal organic disease (i.e. celiac disease, inflammatory bowel diseases).

E 03. A positive diagnosis of irritable bowel syndrome based on the Rome IV criteria questionnaire which requires the patient to experience abdominal pain at least weekly

E 04. Reported history of previous major abdominal surgery (excluding appendectomy and cholecystectomy)

E 05. Any medical condition making participation potentially compromising the participation in the study (e.g. diabetes mellitus, respiratory disease limiting ability to lie in the scanner, known allergy to one of the food products) as per investigator's judgment

E 06. Contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury

E 07. Any condition incompatible with the patient's participation to the study as per investigator's judgment.

E 08. Not willing or able agree to dietary restrictions required in 24 hours before each MRI study day

E 09. Anticipate need for antibiotics intake during the study.

E 10. Unwilling to stop probiotics for the duration of the study period

E 11. Unable/ not willing to stop drugs known to alter GI motility including, regular loperamide, antispasmodics, (e.g. buscopan, mebeverine, peppermint oil, alverine citrate), eluxadoline opiates, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists for the duration of the study (Selective serotonin reuptake inhibitors and low dose tricyclic antidepressants (< 30mg amitriptyline or 50mg nortriptyline) will be recorded but provided dose is stable, will not be an exclusion criteria).

E 12. Having taken part in a research study within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Consistency of chyme in ascending colon | Area under the curve 300-450 minutes after single intake of intervention
  as measured by MRI (T1)

SECONDARY OUTCOMES:
Longer term consistency of chyme in ascending colon | 24 hours after drug intake
  as measured by MRI (T1)
Gut motor function | 0-150 and 150-450 minutes after single intake of intervention
  colonic and small bowel motility as measured by MRI
Small intestinal water content | 0-150 and 150-450 minutes after single intake of intervention
  as measured by MRI
Colon volumes | 0-150 and 150-450 minutes after single intake of intervention
  as measured by MRI
Speed of whole gut transit | at 450 minutes and 24 hours after transit marker and study drug intake
  weighted average position score of transit markers

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
For those journals that request sharing of the analyzable data sets that are reported in the publication, interested researchers are directed to submit their request to clinicalstudydatarequest.com.